CLINICAL TRIAL: NCT02807415
Title: Intestinal Current Measurements (ICM) to Evaluate the Activation of Mutant CFTR in Subjects With Cystic Fibrosis Aged 12 Years and Older, Homozygous for the p.Phe508del-CFTR Mutation, Treated With Lumacaftor in Combination With Ivacaftor
Brief Title: ICM to Evaluate the Activation of p.Phe508del-CFTR by Lumacaftor in Combination With Ivacaftor
Acronym: OrkambiFacts
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Heidelberg University (Other); University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: 2846-2015 82DZLE12A1
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; CFTR; CFTR modulation; sweat test; intestinal current measurement, ICM; nasal transepithelial potential difference measurement, NPD
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor; lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lumacaftor plus Ivacaftor — Oral treatment with lumacaftor/ivacaftor tablets according to the prescribing information
  Other Names: Orkambi; VX-770; VX-809

SUMMARY:
The academic investigator - initiated trial will evaluate in a postapproval setting whether, and if yes, to what extent and variability, the treatment with lumacaftor in combination with ivacaftor reverses the p.Phe508del CFTR - mediated basic defect in p.Phe508del homozygous subjects with cystic fibrosis under real life conditions.

DETAILED DESCRIPTION:
Study design. This academic investigator - initiated trial will resolve the key issue whether, and if yes, to what extent and variability, the treatment with lumacaftor in combination with ivacaftor (Orkambi®) will reverse the p.Phe508del CFTR - mediated basic defect in p.Phe508del homozygous subjects with cystic fibrosis (CF) under real life conditions.

Each p.Phe508del homozygous subject will function as his own control. Baseline measurements will be performed within a 4-week interval prior to the start of oral treatment with lumacaftor + ivacaftor. According to the phase 3 study results by week 4 the gain of FEV1 levels off, drug levels are in steady state and all reversible initial reductions of lung function are resolved. Thus the second assessment will be performed during the initial steady state at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor + ivacaftor. At both days of investigations the basic defect will be assessed by Gibson-Cooke pilocarpine iontophoresis sweat test, nasal transepithelial potential difference measurement (NPD) and intestinal current measurement (ICM). Moreover lung function will be measured by spirometry. The plasma concentrations of lumacaftor, ivacaftor, and their metabolites will be determined and the safety of the oral treatment with Orkambi will be assessed according to the prescribing information.

Study participants will be requested to record the administration of Orkambi® by date and time for 7 days before the scheduled visit to perform functional CFTR assays. Orkambi® should be administered within 30 minutes of consuming fat-containing food according to the FDA-approved patient labeling and the prescribing information. Subjects will be given a diary to record the time and doses of administration of Orkambi® for seven days before the scheduled visit.

Measures against recruitment bias. The local patient databases at the three sites will be searched for all subjects who fulfil the inclusion criteria. After all subjects have been removed from the list who fulfill one or more exclusion criteria, the eligible subjects will be randomly assigned to rank numbers. Subjects will then be contacted in the sequence as they appear in the rank number list.

Statistical analysis. The sample size estimate is based on the absolute change from baseline of the cumulative chloride secretory ion current response to forskolin/Isobutyl methyl xanthine (IBMX) and carbachol in ICM as outcome measure of CFTR function. Assuming a nominal type I error of 0.05 and a power of 0.8, 125 or 33 subjects are needed to demonstrate a treatment effect of 5% or 10%, respectively. Thus even modest changes in the basis defect can be demonstrated in a recruited cohort of 125 subjects and incomplete data sets in up to half of all subjects.

To evaluate changes in lung function and CFTR biomarkers prior and during treatment with Orkambi® , Student's t test, paired Student's t test or Wilcoxon signed-rank test will be performed as appropriate. Relationships between CFTR biomarkers will be first assessed by the Pearson product-moment correlation coefficient and in case that the whole data set will be explored by canonical correlation analysis. Furthermore the sensitivity and specificity of the CFTR biomarkers in detecting treatment effects will be determined. The biostatistician from the Koordinierungszentrum für Klinische Studien (KKS) Heidelberg will assist in the statistical evaluation.

Ethical considerations. Orkambi® has been approved for treatment of subjects with cystic fibrosis, homozygous for the p.Phe508del mutation. Drug handling and safety controls will be executed according to the Bundesinstitut für Arzneimittel und Medizinprodukte (BfArM)-approved patient labeling and full prescribing information.

Study protocol and informed consent forms were approved by the ethics committees. Prior to any investigation patients and their parental guides (if applicable) will be informed about the background, objectives, schedule and assessments of the study. Each adult aged 18 years or older must sign and date the study-specific informed-consent form before any study-specific procedures can be performed. Subjects aged 12 - 17 years must assent to participate in the study and the subject's parent or legal guardian must sign and date the study-specific informed-consent form before any study-specific procedures can be performed.

Sweat test and NPD are safe procedures. Burns during iontophoresis, injuries by placement of the subcutaneous electrode for NPD or diuresis induced by swallowing of amiloride in younger subjects during nasal superfusion have not been observed at the three sites.

The collection of rectal biopsies is principally a safe and painless procedure. ICM has been performed at Hannover Medical School. since 1995. During these 20 years bleedings have been observed in five subjects one of whom required hospitalization. Haemorrhoids and abnormal bleeding times are contraindications for ICM and are exclusion criteria to participate in the study. Hence, with the exception of the low bleeding risk associated with the collection of rectal biopsies study participants are not put at risk.

There is no direct benefit for study participants, however, the decision whether or not Orkambi® should be prescribed can be based on solid data.

Quality assurance. Sweat test, NPD, ICM and sampling (blood, serum, plasma) will be performed according to harmonized Standard Operating Procedures based on protocols of the Clinical Trials Network of the European Cystic Fibrosis Society and/or the Therapeutics Development Network Coordinating Center of the US Cystic Fibrosis Foundation and/or the Hannover Unified Biobank. Pre-study hands-on meetings have been organized to compare on-site the execution of the protocols including sweat test, NPD, ICM, lung function testing and sampling, processing, storage of serum and plasma specimens. Sweat testing is subject to domestic quality control trials. Local and central reading will be performed for all NPD and ICM tracings. The sites have long-standing expertise in CFTR biomarkers and have trained numerous domestic and European sites in NPD and ICM. - Subjects will be educated in drug dosing. A diary with drug dosing (date and time) will be filled out during the 7 days prior to the day of assessment.

ELIGIBILITY:
Inclusion Criteria:

1. p.Phe508del homozygous subjects aged 6 years and older with cystic fibrosis
2. FEV1 ≥ 40% of predicted normal for age, gender and height (Knudson standards) or FEV1 > 35% of predicted normal for age, gender and height at baseline, stable lung function during the preceding three months and no acute upper or lower respiratory infection or pulmonary exacerbation during the preceding four weeks
3. Hematology, serum chemistry, coagulation results at baseline with no clinically significant abnormalities that would interfere with the oral treatment with Orkambi® and with the study assessments, as judged by the investigator
4. Able to understand and comply with protocol requirements, restrictions, and instructions and likely to complete the study as planned, as judged by the investigator
5. Willing to remain on a stable medication regimen and administration of Orkambi® according to the FDA-approved patient labeling and the prescribing information for the duration of study participation -

Exclusion Criteria:

1. History of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering Orkambi®
2. An acute upper or lower respiratory infection or pulmonary exacerbation at baseline
3. Advanced liver disease as documented by sonography
4. Abnormal liver function at baseline, defined as ≥ 3 upper limit of normal in minimum 3 of the following: serum aspartate transaminase, serum alanine transaminase, gamma-glutamyl transpeptidase, or total bilirubin
5. Abnormal blood creatine phosphokinase at baseline
6. Abnormal renal function at baseline, defined as creatinine clearance < 60 mL/min
7. Co-medication with strong Cytochrome P450, Family 3, subfamily A (CYP3A) inhibitors and inducers
8. Non-congenital lens opacities
9. Haemorrhoids (bleeding risk when taking rectal suction biopsies for ICM)
10. History of nasal surgery that removed the respiratory epithelium
11. Topical treatment of nostrils in the 3 days prior to baseline
12. Disturbing nasal aspects of secretions, erythema, crustae, ulcera, edema at baseline
13. Participation in a clinical study involving administration of a CFTR modulator
14. History of solid organ or haematological transplantation
15. History of alcohol, medication, or illicit drug abuse Exclusion criteria 1, 3, 4, 5, 6, 7 and 8 refer to known risk factors for the treatment with Orkambi®.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with cystic fibrosis aged 6 years and older, homozygous for the p.Phe508del-CFTR mutation
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
ICM Absolute change from baseline of the cumulative chloride secretory ion current response to forskolin/IBMX and carbachol in rectal tissue as a CFTR biomarker | Measurement at the baseline visit within a 4-week interval prior to the start of oral treatment with lumacaftor and ivacaftor; second measurement at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor and ivacaftor
  ICM will be performed according to the Standard Operating Procedure ICM_EU001, version 2.7 (October 2011) 'Ion Transport in Rectal Biopsies for Diagnosis and Clinical Trials in Cystic Fibrosis of the European Cystic Fibrosis Society (ECFS) Diagnostic Working Group & Clinical Trials Network modified by in-house protocol adjustments at the CF electrophysiology laboratories in Hannover and Heidelberg as described by Graeber et al. (2015) [39]. Electronic files of the tracings will be evaluated on-site and at the CF Electrophysiology Laboratory at the University of Heidelberg.

SECONDARY OUTCOMES:
Spirometry Absolute change from baseline in percent predicted forced expiratory volume in 1 second (FEV1) | Measurement at the baseline visit within a 4-week interval prior to the start of oral treatment with lumacaftor and ivacaftor; second measurement at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor and ivacaftor
  Pre-bronchodilator spirometry will be performed using in-house equipment. Pre-bronchodilator spirometry is defined as spirometry testing performed for a subject who has
  * Withheld short-acting bronchodilators or anticholinergic agents for more than 4 hours before the spirometry assessment; and
  * Withheld their long-acting bronchodilator (e.g., salmeterol) more than 12 hours before the spirometry assessment; and
  * Withheld their once-daily, long-acting bronchodilator (e.g., tiotropium bromide) for more than 24 hours before the spirometry assessment.
NPD Absolute change from baseline of the Sermet score of nasal transepithelial potential difference measurements (NPD) as a CFTR biomarker | Measurement at the baseline visit within a 4-week interval prior to the start of oral treatment with lumacaftor and ivacaftor; second measurement at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor and ivacaftor
  NPD will be performed according to the Standard Operating Procedure NPD_EU001, version 1.7 (March 2013) 'Nasal Potential Difference (NPD) Measurement for Diagnosis and Clinical Trials in Cystic Fibrosis' of the European Cystic Fibrosis Society (ECFS) Diagnostic Working Group & Clinical Trials Network. Electronic files of the tracings will be evaluated on-site and at the CF Electrophysiology Laboratory of Hannover Medical School.
Sweat chloride testing Absolute change from baseline of the chloride concentration in Gibson-Cooke pilocarpine iontophoresis sweat test as a CFTR biomarker | Measurement at the baseline visit within a 4-week interval prior to the start of oral treatment with lumacaftor and ivacaftor; second measurement at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor and ivacaftor
  The sweat test will be performed according the Clinical and Laboratory Standards Institute guidelines (Clinical and Laboratory Standards Institute: Sweat Testing: Sample Collection and Quantitative Chloride Analysis; Approved Guideline-Third Edition, document C34-A3. Wayne, PA, USA: Clinical and Laboratory Standards Institute; 2009). After stimulation of sweat production by pilocarpine iontophoresis and collection of sweat (Macroduct®; Wescor Inc., Logan, NV, USA), the sweat chloride concentration is determined in-house by original titration with a chloridometer.

OTHER OUTCOMES:
Drug testing Plasma concentrations of lumacaftor, ivacaftor, and their metabolites | Measurement at the baseline visit within a 4-week interval prior to the start of oral treatment with lumacaftor and ivacaftor; second measurement at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor and ivacaftor
  Whole blood samples will be collected. Plasma will be assayed by high-performance liquid chromatography.
Safety Issues assessed by Liver-related events, respiratory events and elevation of blood creatine phosphokinase | Measurement at the baseline visit within a 4-week interval prior to the start of oral treatment with lumacaftor and ivacaftor; second measurement at a day 10 - 14 weeks after the initiation of oral treatment with lumacaftor and ivacaftor
  Liver-related events (serum serum aspartate transaminase, serum alanine transaminase, gamma-glutamyl transpeptidase, total bilirubin), respiratory events (chest discomfort, dyspnea, and respiration abnormal) and elevation of blood creatine phosphokinase will be monitored according to the FDA-approved patient labeling and the prescribing information.

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Tümmler, MD PhD, Principal Investigator — Hannover Medical School; Marcus Mall, MD, Principal Investigator — Heidelberg University; Lutz Nährlich, MD, Principal Investigator — University of Giessen
Locations (3):
- Germany (3):
  - Justus-Liebig-University, Giessen
  - Hannover Medical School, Hanover
  - University of Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to study participant and parental guide and the physician treating the study participant
Supporting Information: Study Protocol, ICF
Time Frame: IPD data are made available in a written summary report to the physician treating the study participant within 4 weeks after study day 2
Access Criteria: access criterion: - the individual study participant gains access to printouts of sweat chloride concentration, NPD and ICM tracings upon request.
  - the physician treating the study participant receives a written report for this subject that summarizes the findings of spirometry, sweat chloride concentration, NPD and ICM tracings.

REFERENCES:
- [Background] Wainwright CE, Elborn JS, Ramsey BW, Marigowda G, Huang X, Cipolli M, Colombo C, Davies JC, De Boeck K, Flume PA, Konstan MW, McColley SA, McCoy K, McKone EF, Munck A, Ratjen F, Rowe SM, Waltz D, Boyle MP; TRAFFIC Study Group; TRANSPORT Study Group. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Jul 16;373(3):220-31. doi: 10.1056/NEJMoa1409547. Epub 2015 May 17. PMID 25981758
- [Background] Elborn JS, Ramsey BW, Boyle MP, Konstan MW, Huang X, Marigowda G, Waltz D, Wainwright CE; VX-809 TRAFFIC and TRANSPORT study groups. Efficacy and safety of lumacaftor/ivacaftor combination therapy in patients with cystic fibrosis homozygous for Phe508del CFTR by pulmonary function subgroup: a pooled analysis. Lancet Respir Med. 2016 Aug;4(8):617-626. doi: 10.1016/S2213-2600(16)30121-7. Epub 2016 Jun 10. PMID 27298017
- [Background] Graeber SY, Hug MJ, Sommerburg O, Hirtz S, Hentschel J, Heinzmann A, Dopfer C, Schulz A, Mainz JG, Tummler B, Mall MA. Intestinal Current Measurements Detect Activation of Mutant CFTR in Patients with Cystic Fibrosis with the G551D Mutation Treated with Ivacaftor. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1252-5. doi: 10.1164/rccm.201507-1271LE. No abstract available. PMID 26568242
- [Result] Graeber SY, Dopfer C, Naehrlich L, Gyulumyan L, Scheuermann H, Hirtz S, Wege S, Mairbaurl H, Dorda M, Hyde R, Bagheri-Hanson A, Rueckes-Nilges C, Fischer S, Mall MA, Tummler B. Effects of Lumacaftor-Ivacaftor Therapy on Cystic Fibrosis Transmembrane Conductance Regulator Function in Phe508del Homozygous Patients with Cystic Fibrosis. Am J Respir Crit Care Med. 2018 Jun 1;197(11):1433-1442. doi: 10.1164/rccm.201710-1983OC. PMID 29327948
- [Derived] Graeber SY, Boutin S, Wielputz MO, Joachim C, Frey DL, Wege S, Sommerburg O, Kauczor HU, Stahl M, Dalpke AH, Mall MA. Effects of Lumacaftor-Ivacaftor on Lung Clearance Index, Magnetic Resonance Imaging, and Airway Microbiome in Phe508del Homozygous Patients with Cystic Fibrosis. Ann Am Thorac Soc. 2021 Jun;18(6):971-980. doi: 10.1513/AnnalsATS.202008-1054OC. PMID 33600745